CLINICAL TRIAL: NCT04740970
Title: A Phase 2a, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Proof of Concept Study to Evaluate the Efficacy, Safety, and Tolerability of JNJ-64304500 in Patients With Alopecia Areata
Brief Title: A Study of JNJ-64304500 in Participants With Alopecia Areata
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108941; 2020-004500-34 (EudraCT Number); 64304500ALA2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-02-03; First posted 2021-02-05 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- JNJ-64304500 (Experimental): Participants will receive JNJ-64304500 dose 1 subcutaneous (SC) injection at Week 0 and then dose 2 SC injection every 2 weeks from Week 2 through Week 22.
  Interventions: Drug: JNJ-64304500
- Placebo (Placebo Comparator): Participants will receive matching placebo SC injection at Week 0 and then every 2 weeks from Week 2 through Week 22.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-64304500 — JNJ-64304500 injection will be administered subcutaneously.
  Arms: JNJ-64304500
Drug: Placebo — Matching placebo injection will be administered subcutaneously.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the clinical response of 22 weeks of study intervention with JNJ-64304500, compared with placebo, in participants with moderate to severe alopecia areata (AA).

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has a physician confirmed diagnosis of moderate to severe Alopecia Areata (AA) (greater than or equal to [>=] 50 percent [%] scalp involvement) as measured using the severity of Alopecia tool (SALT) score; or participant has >=95% loss of scalp hair for enrollment as alopecia totalis (AT) or alopecia universalis (AU) subtypes at the time of screening and baseline
* Current episode of hair loss is greater than (>) 6 months (without evidence of spontaneous terminal hair regrowth within 6 months at the time of screening and baseline), but less than or equal to (<=8) years
* Medically stable on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at either screening or Week 0. Any abnormalities, must be consistent with the underlying illness in the study population and this determination must be recorded in the participant's source documents and initialed by the investigator
* Medically stable on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel or hematology are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator

Key Exclusion Criteria:

* History of liver or renal insufficiency (estimated creatinine clearance below 60 milliliters per minute (mL/min)); significant cardiac, vascular, pulmonary, gastrointestinal, endocrine (except stable thyroid diseases), neurologic, hematologic, rheumatologic, psychiatric disorders, or metabolic disturbances
* Currently has a malignancy or has a history of malignancy (with the exceptions of participants having adequately treated and cured basal or squamous cell carcinoma of the skin, or cervical carcinoma in situ occurring more than 5 years prior to randomization)
* Known allergies, hypersensitivity, or intolerance to JNJ-64304500 or its excipients
* Participants with current episode of hair loss for >8 years
* Has previous treatment with an oral janus kinase (JAK) inhibitor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-24 (Estimated); Primary Completion 2022-06-02 (Estimated); Study Completion 2022-07-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a Severity of Alopecia Tool (SALT)90 Response | Week 24
  The SALT score is a global severity score that captures percentage of hair loss by dividing the scalp into 4 quadrants (left side, right side, top and back quadrant) with assigned percent of scalp surface area (SSA) in each quadrant. After indicating the percent of loss per quadrant the value is multiplied by the percent (%) of hair for each section (18% sides, 40% top, and 24% back) and the values are summed to generate the total percentage of scalp hair loss or SALT score. The range in score is from 0-100 reflecting the percent hair loss on the scalp (0=no hair loss and 100= total hair loss). SALT90 is defined as 90% or more regrowth compared with baseline.

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Up to Weeks 24 and 38
  Number of participants with TEAEs will be reported. An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants With Treatment-emergent Serious Adverse Events (SAEs) | Up to Weeks 24 and 38
  Number of participants with treatment-emergent SAEs will be reported. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Number of Participants With Adverse Events Leading to Discontinuation of Study Intervention | Up to Weeks 24 and 38
  Number of participants with AEs leading to discontinuation of study will be reported.
Number of Participants With Adverse Events Reasonably Related to Study Intervention | Up to Weeks 24 and 38
  Number of participants with AEs reasonably related to study intervention will be reported.
Number of Participants With Adverse Events of Injection-Site Reactions | Up to Weeks 24 and 38
  Number of participants with AEs of injection-site reactions will be reported. An injection-site reaction is any AE at a subcutaneous (SC) study intervention injection-site.
Number of Participants with Adverse Events of Infections | Up to Weeks 24 and 38
  Number of participants with AEs of infections, including serious infections (including reactivation of latent infections) and infections requiring oral or parenteral antimicrobial treatment will be reported.
Number of Participants With Clinically Significant Abnormalities in Vital Signs | Up to Weeks 24 and 38
  Number of participants with clinically significant abnormalities in vital signs including pulse rate, respiratory rate and blood pressure will be reported.
Number of Participants With Clinically Significant Abnormalities in Laboratory Tests | Up to Weeks 24 and 38
  Number of participants with clinically significant abnormalities in laboratory tests including hematology and chemistry will be reported.
Percentage of Participants Achieving SALT50 Response | Week 24
  Percentage of participants achieving SALT50 response will be reported. The SALT score is a global severity score that captures percentage of hair loss by dividing the scalp into 4 quadrants (left side, right side, top and back quadrant) with assigned percent of SSA in each quadrant. After indicating the percent of loss per quadrant the value is multiplied by the percent of hair for each section (18% sides, 40% top, and 24% back) and the values are summed to generate the total percentage of scalp hair loss or SALT score. The range in score is from 0-100 reflecting the percent hair loss on the scalp (0=no hair loss and 100= total hair loss). SALT50 is defined as 50% or more regrowth from baseline.
Percentage of Participants Achieving SALT75 Response | Week 24
  Percentage of participants achieving SALT75 response will be reported. The SALT score is a global severity score that captures percentage of hair loss by dividing the scalp into 4 quadrants (left side, right side, top and back quadrant) with assigned percent of SSA in each quadrant. After indicating the percent of loss per quadrant the value is multiplied by the percent of hair for each section (18% sides, 40% top, and 24% back) and the values are summed to generate the total percentage of scalp hair loss or SALT score. The range in score is from 0-100 reflecting the percent hair loss on the scalp (0=no hair loss and 100= total hair loss). SALT75 is defined as 75% or more regrowth from baseline.
Change From Baseline in SALT Score at Week 24 | Baseline and Week 24
  Change from baseline in SALT score at Week 24 will be reported. The SALT score is a global severity score that captures percentage of hair loss by dividing the scalp into 4 quadrants (left side, right side, top and back quadrant) with assigned percent of SSA in each quadrant. After indicating the percent of loss per quadrant the value is multiplied by the percent of hair for each section (18% sides, 40% top, and 24% back) and the values are summed to generate the total percentage of scalp hair loss or SALT score. The range in score is from 0-100 reflecting the percent hair loss on the scalp (0=no hair loss and 100= total hair loss).
Percent Change in SALT Score from Baseline at Week 24 | Baseline and Week 24
  Percent change from baseline in SALT score at Week 24 will be reported. The SALT score is a global severity score that captures percentage of hair loss by dividing the scalp into 4 quadrants (left side, right side, top and back quadrant) with assigned percent of SSA in each quadrant. After indicating the percent of loss per quadrant the value is multiplied by the percent of hair for each section (18% sides, 40% top, and 24% back) and the values are summed to generate the total percentage of scalp hair loss or SALT score. The range in score is from 0-100 reflecting the percent hair loss on the scalp (0=no hair loss and 100= total hair loss).
Percentage of Participants Achieving SALT Score Less Than or Equal to (<=) 10 | Week 24
  Percentage of participants with SALT score <=10 will be reported. The SALT score is a global severity score that captures percentage of hair loss by dividing the scalp into 4 quadrants (left side, right side, top and back quadrant) with assigned percent of SSA in each quadrant. After indicating the percent of loss per quadrant the value is multiplied by the percent of hair for each section (18% sides, 40% top, and 24% back) and the values are summed to generate the total percentage of scalp hair loss or SALT score. The range in score is from 0-100 reflecting the percent hair loss on the scalp (0=no hair loss and 100= total hair loss).
Percentage of Participants Achieving SALT Score <=20 | Week 24
  Percentage of participants with SALT score <=20 will be reported. The SALT score is a global severity score that captures percentage of hair loss by dividing the scalp into 4 quadrants (left side, right side, top and back quadrant) with assigned percent of SSA in each quadrant. After indicating the percent of loss per quadrant the value is multiplied by the percent of hair for each section (18% sides, 40% top, and 24% back) and the values are summed to generate the total percentage of scalp hair loss or SALT score. The range in score is from 0-100 reflecting the percent hair loss on the scalp (0=no hair loss and 100= total hair loss).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (22):
- United States (9):
  - Forcare Clinical Research, Inc., Tampa, Florida
  - Indiana Clinical Trial Center, Plainfield, Indiana
  - Dermatology Specialists, Louisville, Kentucky
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Oregon Dermatology and Research Center, Portland, Oregon
  - University of Pittsburgh Department of Dermatology, Pittsburgh, Pennsylvania
  - Modern Research Associates, Dallas, Texas
  - Center for Clinical Studies, Webster, Texas
- Australia (4):
  - Sinclair Dermatology, East Melbourne
  - Fremantle Dermatology, Fremantle
  - St George Dermatology & Skin Cancer Centre, Kogarah
  - Veracity Clinical Research, Woolloongabba
- France (3):
  - CHU Bordeaux - Hopital St Andre, Bordeaux
  - CHU de Nice Hopital de l Archet, Nice
  - CHU Rouen - Hopital Charles Nicolle, Rouen
- Japan (6):
  - Hamamatsu University Hospital, Hamamatsu
  - Kyorin University Hospital, Mitaka
  - Osaka City University Hospital, Osaka
  - The Juntendo Tokyo Koto Geriatric Medical Center, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Yamaguchi University Hospital, Ube

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency